CLINICAL TRIAL: NCT02844036
Title: Angioplasty of Distal Lesions for Carriers of Inoperable Post-embolic HTP
Acronym: OCT²EPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC13.440
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Hypertension
Keywords: Distal Lesions; Post-embolic HTP; Angioplasty
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with a pulmonary hypertension (Experimental): Pulmonary hypertension group 4 of Dana point, chronic thromboses lesions, thromboembolic.
  Interventions: Procedure: Percutaneous angioplasty; Procedure: Balloon angioplasty; Procedure: Right heart catheterization; Procedure: Echocardiography; Other: A six-minute walking test; Procedure: Functional respiratory investigations; Procedure: Pulmonary tomography or pulmonary angiography; Other: Biological parameters

INTERVENTIONS:
Procedure: Percutaneous angioplasty
Procedure: Balloon angioplasty
Procedure: Right heart catheterization
Procedure: Echocardiography
Other: A six-minute walking test
Procedure: Functional respiratory investigations
Procedure: Pulmonary tomography or pulmonary angiography
Other: Biological parameters

SUMMARY:
Currently, the standard treatment for proximal thromboses lesions responsible for post-embolic pulmonary hypertension, is the surgical thromboendarterectomy. When the ravages are judged too distal or the patient is judged inoperable for a curative surgical gesture, there is no evidence of any therapeutic option, exept for K anti-vitamins for recurrent embolism. Prognosis is then pejorative with a 60% mortality at 5 years.

This study propose an alternative treatment for these patients in therapeutic "dead end". This is about applying arterial thrombosis technique to the pulmonary circulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients with a pulmonary hypertension diagnosed by right catheterisation, with a mean arterial pressure >30 mmHg and arterial pulmonary resistance > 3 UW.
* Patients with group 4 (Dana point) pulmonary hypertension, thromboembolic.
* Chronic thrombosis visible to scanner, pulmonary IRM angiogram or to pulmonary angiogram.
* Patient's file refused by the reference center multidisciplinary coordination meetings for surgical thromboendartériectomy or refusal from the patient to be operate.
* Absence of counter-argument to the femoral venous or jugular way.
* Normal kidney function or moderatly degraded (clearance>30 mL) or dialysed renal failure
* Persons affiliated to national social security
* Signed free consent by patients

Exclusion Criteria:

* Pulmonary hypertension pos-embolic operated by thromboendarteriectomy
* Pulmonary hypertension Group 1 of Dana Point, meaning idiopathic, familial, post-anorectics, associate with a congenital heart disease associated to a scleroderma, associated to a chronic hemolytic disease
* Pulmonary hypertension Group 2 of Dana Point, associated with a left cardiovascular disease
* Pulmonary hypertension Group 3 of Dana Point, associated to a respiratory disease
* Pulmonary hypertension Group 5 of Dana Point, of unclear or multifactorial mechanism
* Hypersensitivity to HEXABRIX, to iodinated contrast product or one of its components
* Obvious thyrotoxicosis
* Protected major persons
* Pregnant or breastfeeding women
* Persons deprived of liberty
* Persons in emergency situations.
* No consent signed or approoved
* Persons no affiliated to national social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Percutaneous angioplasty | About 90 minutes
  International Normalized Ratio wil be measure and need to be between 2 and 3.
Balloon angioplasty | About 90 minutes
  Same mode than valscular or coronal angioplasty.
Right heart catheterization | Few minutes
  Right auricular pressure auriculaire droite moyenne ou POD (mmHg)
  * Blood pressure : systolic, diastolic, and average(mmHg)
  * pression artérielle pulmonaire d'occlusion (PAPO) moyenne (mmHg)
Echocardiography | Few minutes
  Right ventricular heart function with evaluation of :
  - The maximum pressure gradient (mmHg)
Walking test | 6 minutes
  Start heart rate (T0) and at the end (T6) of the test (bpm)
Functional respiratory investigations | About an hour
  * Forced expiratory volume (FEV) ml/kg
  * Forced vital capacity (FVC) ml/kg
  * Total lung capacity ml/kg
  * Alveolar capillarytransfer of Carbon monoxide (CO) ml/kg
  * Transfer coefficient of CO (KCO) ml/kg
  All volumes in ml/kg
Pulmonary tomography or pulmonary angiography | About 30 minutes
  tomography (CT) or angiography
Heart rate | Few minutes
  Heart rate (bpm) during right heart catheterization.
Cardiac output (L/min) | Few minutes
  Cardiac output (L/min) during right heart catheterization.
Venous oxygen saturation (%) | Few minutes
  Venous oxygen saturation (%) during right heart catheterization.
Echocardiography | Few minutes
  Right ventricular heart function with evaluation of :
  Surface area of the right ventricle (cm²)
Echocardiography | Few minutes
  Right ventricular heart function with evaluation of :
  Cardiac output (L/min) and cardiac index (L/min/m²)
Walking test | 6 minutes
  Patient self evaluation of the dyspnea on a Borg scale from 0 (not breathless) to 10 (serious breathless)
Walking test | 6 minutes
  Arterial blood saturation in oxygen measured by an oxymeter dat the beginning (T0) and at the end of the test (T6) (SO2)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Bouvaist, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Mizoguchi H, Ogawa A, Munemasa M, Mikouchi H, Ito H, Matsubara H. Refined balloon pulmonary angioplasty for inoperable patients with chronic thromboembolic pulmonary hypertension. Circ Cardiovasc Interv. 2012 Dec;5(6):748-55. doi: 10.1161/CIRCINTERVENTIONS.112.971077. Epub 2012 Nov 27. PMID 23192917
- [Background] Sugimura K, Fukumoto Y, Satoh K, Nochioka K, Miura Y, Aoki T, Tatebe S, Miyamichi-Yamamoto S, Shimokawa H. Percutaneous transluminal pulmonary angioplasty markedly improves pulmonary hemodynamics and long-term prognosis in patients with chronic thromboembolic pulmonary hypertension. Circ J. 2012;76(2):485-8. doi: 10.1253/circj.cj-11-1217. Epub 2011 Dec 15. PMID 22185711
- [Background] Fukumoto Y, Shimokawa H. Recent progress in the management of pulmonary hypertension. Circ J. 2011;75(8):1801-10. doi: 10.1253/circj.cj-11-0567. Epub 2011 Jul 11. PMID 21747194
- [Background] Feinstein JA, Goldhaber SZ, Lock JE, Ferndandes SM, Landzberg MJ. Balloon pulmonary angioplasty for treatment of chronic thromboembolic pulmonary hypertension. Circulation. 2001 Jan 2;103(1):10-3. doi: 10.1161/01.cir.103.1.10. PMID 11136677
- [Background] Jais X, D'Armini AM, Jansa P, Torbicki A, Delcroix M, Ghofrani HA, Hoeper MM, Lang IM, Mayer E, Pepke-Zaba J, Perchenet L, Morganti A, Simonneau G, Rubin LJ; Bosentan Effects in iNopErable Forms of chronIc Thromboembolic pulmonary hypertension Study Group. Bosentan for treatment of inoperable chronic thromboembolic pulmonary hypertension: BENEFiT (Bosentan Effects in iNopErable Forms of chronIc Thromboembolic pulmonary hypertension), a randomized, placebo-controlled trial. J Am Coll Cardiol. 2008 Dec 16;52(25):2127-34. doi: 10.1016/j.jacc.2008.08.059. PMID 19095129
- [Background] Diggle PJ, Liang KY, Zeger SL. Analysis of longitudinal data. New York: Oxfiord University Press, 2000.
- [Background] Twisk JWR. Applied longitudinal analysis for epidemiology. Cambridge: Cambridge University Press, 2003.
- [Background] Mayer E, Jenkins D, Lindner J, D'Armini A, Kloek J, Meyns B, Ilkjaer LB, Klepetko W, Delcroix M, Lang I, Pepke-Zaba J, Simonneau G, Dartevelle P. Surgical management and outcome of patients with chronic thromboembolic pulmonary hypertension: results from an international prospective registry. J Thorac Cardiovasc Surg. 2011 Mar;141(3):702-10. doi: 10.1016/j.jtcvs.2010.11.024. PMID 21335128
- [Background] Pepke-Zaba J, Jansa P, Kim NH, Naeije R, Simonneau G. Chronic thromboembolic pulmonary hypertension: role of medical therapy. Eur Respir J. 2013 Apr;41(4):985-90. doi: 10.1183/09031936.00201612. Epub 2013 Feb 8. PMID 23397304
- [Background] de Perrot M, McRae K, Shargall Y, Pletsch L, Tan K, Slinger P, Ma M, Paul N, Moric J, Thenganatt J, Mak S, Granton JT. Pulmonary endarterectomy for chronic thromboembolic pulmonary hypertension: the Toronto experience. Can J Cardiol. 2011 Nov-Dec;27(6):692-7. doi: 10.1016/j.cjca.2011.09.009. Epub 2011 Oct 21. PMID 22018451
- [Background] Inami T, Kataoka M, Shimura N, Ishiguro H, Yanagisawa R, Taguchi H, Fukuda K, Yoshino H, Satoh T. Pulmonary edema predictive scoring index (PEPSI), a new index to predict risk of reperfusion pulmonary edema and improvement of hemodynamics in percutaneous transluminal pulmonary angioplasty. JACC Cardiovasc Interv. 2013 Jul;6(7):725-36. doi: 10.1016/j.jcin.2013.03.009. Epub 2013 Jun 14. PMID 23769649